CLINICAL TRIAL: NCT01094236
Title: Interactive Program for Effective Playground Supervision
Acronym: Playground_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Responsible Party: Lynne H. Grilley Swartz, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SBIR40-2
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Behavior
Keywords: behavior management; academic performance; playground supervision; harm reduction; Behavioral Research
MeSH Terms: conditions — Behavior; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Supervisor Treatment Group (Experimental): Supervisors watched the CD intervention
  Interventions: Behavioral: On the Playground behavior management program
- Administrators - Treatment (Experimental): School administrators got access to the intervention binder with CD's, workbook and worksheets
  Interventions: Behavioral: On the Playground behavior management program
- Students (Experimental): 3rd grade students at participating study schools
  Interventions: Behavioral: On the Playground behavior management program
- Supervisor Control Group (Experimental): Supervisors watched a video on playground equipment safety
  Interventions: Behavioral: On the Playground behavior management program
- Administrators - Control (Experimental): Administrators did not have access to any treatment materials.
  Interventions: Behavioral: On the Playground behavior management program
- School Staff (Experimental): School staff surveyed at staff meetings
  Interventions: Behavioral: On the Playground behavior management program

INTERVENTIONS:
Behavioral: On the Playground behavior management program — Treatment school playground supervisors were show the CD intervention. Control school playground supervisors were given a video on playground equipment safety. All school staff subjects were assessed before the intervention and 75 days following the supervisor intervention. Students were assessed before the intervention, and then 45 days and 75 days following the supervisor intervention. School Administrators were assessed before the intervention, and then 30 and 60 days after the supervisor intervention - school administrators at treatment schools had access to a treatment binder with CDs and worksheets, while the control school administrators did not.
  Other Names: A Guide to Playground Management

SUMMARY:
The goal of the Playground supervision clinical trial is to see if playground management skills are improved, after implementing the school-wide behavior management program.

DETAILED DESCRIPTION:
The Center for Disease Control and Prevention (CDC) reports that over 200,000 children every year are admitted to emergency rooms due to playground related injuries sustained at school. The National Association for Playground Safety recommends not only improving surface materials and equipment, but also improving adult supervision of children while at play. Yet, there are limited empirical studies in the literature that have examined the impact of a comprehensive training program to improve playground safety by improving supervisor knowledge and attitudes. The purpose of this study was to evaluate the efficacy of a comprehensive, stand-alone interactive multimedia computer-based training program for elementary school faculty to implement a school-wide behavior management program for playground environments. To do this, a randomized control trial comparing the experiences of playground supervisors, students, and staff from schools of a large urban school district was carried out. School was both the unit of randomization and the unit of analysis. The comparisons were measured by pre, post and follow-up assessments conducted by the investigators. Results suggest significant positive differences due to treatment in knowledge, beliefs and attitudes for playground supervisors, students, and staff.

ELIGIBILITY:
Inclusion Criteria:

* school staff in elementary schools (grades K-5)
* must be in the included school district for Las Vegas, NV.

Exclusion Criteria:

* schools outside of the Las Vegas school district
* middle schools
* junior high schools
* high schools

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2316 (Actual)
Dates: Start 2005-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Improved playground management skills for treatment schools | 6 months

SECONDARY OUTCOMES:
Supervisors: Improved knowledge, attitude, intentions and efficacy in implementing effective playground management. | 6 months
Administrators: increased knowledge and attitudes about playground safety when compared to control schools. | 6 months
Students: Increased perception of playground safety compared to control schools | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynne H Grilley Swartz, MPH, CHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States